CLINICAL TRIAL: NCT02373722
Title: Web App Based Patient Education in Mohs Surgery
Brief Title: Website Application Based Education and Text Messaging in Improving Skin Wound Care in Patients Undergoing Mohs Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00028840; NCI-2015-00217 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01714 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Malignant Skin Neoplasm
MeSH Terms: conditions — Skin Neoplasms | interventions — Mohs Surgery; Early Intervention, Educational; Educational Status; Methods; Petrolatum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (video, text message) (Experimental): Patients watch an educational video about Mohs surgery before their surgery, a video about wound care after the surgery and receive text messages about wound care on days 1-5 after the surgery. Patients also receive instructions to reduce movement and use a Fitbit activity tracker. Beginning 48 hours after surgery, patients are instructed to apply petroleum jelly BID to the wound area.
  Interventions: Procedure: Mohs Surgery; Other: Internet-Based Intervention; Behavioral: Telephone-Based Intervention; Other: Educational Intervention; Behavioral: Exercise Intervention; Other: Petrolatum-Mineral Oil-Lanolin-Ceresin Ointment; Other: Questionnaire Administration; Other: Survey Administration
- Group II (educational video) (Experimental): Patients watch an educational video about Mohs surgery before their surgery, an educational video about wound care after the surgery and receive instructions to reduce movement and use a Fitbit activity tracker. Beginning 48 hours after surgery, patients apply petroleum jelly BID to the wound area
  Interventions: Procedure: Mohs Surgery; Other: Internet-Based Intervention; Other: Educational Intervention; Behavioral: Exercise Intervention; Other: Petrolatum-Mineral Oil-Lanolin-Ceresin Ointment; Other: Questionnaire Administration; Other: Survey Administration
- Group III (text message) (Experimental): Patients receive text messages about wound care on days 1-5 after the surgery and receive instructions to reduce movement and use a Fitbit activity tracker. Beginning 48 hours after surgery, patients are also instructed to apply petroleum jelly BID to the wound are.
  Interventions: Procedure: Mohs Surgery; Behavioral: Telephone-Based Intervention; Behavioral: Exercise Intervention; Other: Petrolatum-Mineral Oil-Lanolin-Ceresin Ointment; Other: Questionnaire Administration; Other: Survey Administration
- Group IV (control) (Experimental): Patients receive no video or text messages. Patients receive instructions to reduce movement and use a Fitbit activity tracker. Beginning 48 hours after surgery, patients are also instructed to apply petroleum jelly BID to the wound area.
  Interventions: Procedure: Mohs Surgery; Behavioral: Exercise Intervention; Other: Petrolatum-Mineral Oil-Lanolin-Ceresin Ointment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Procedure: Mohs Surgery — Undergo Mohs surgery
Other: Internet-Based Intervention — Watch website application based educational video
  Arms: Group I (video, text message); Group II (educational video)
Behavioral: Telephone-Based Intervention — Receive text messages
  Arms: Group I (video, text message); Group III (text message)
Other: Educational Intervention — Watch website application based educational video
  Other Names: Education for Intervention; Intervention, Educational
  Arms: Group I (video, text message); Group II (educational video)
Behavioral: Exercise Intervention — Use Fitbit
Other: Petrolatum-Mineral Oil-Lanolin-Ceresin Ointment — Applied to the wound area
  Other Names: Aquaphor
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies how well website application (web app) based education and text messaging works in improving skin wound care in patients undergoing Mohs surgery (a surgical procedure used to treat skin cancer). Website application and text messaging based education may help patients stick to wound care instructions before and after surgery, lower anxiety level, and may help monitor their activity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To create a web application which will educate dermatologic surgery patients prior to their operations with educational videos.

SECONDARY OBJECTIVES:

I. To create and evaluate a web based system to send wound care instructions to patients by text message after their operation.

II. Qualitative comments from participants and research staff concerning the feasibility of this approach and the use of Fitbit activity trackers as a means to monitor movement restriction.

III. The rate of adverse events.

OUTLINE: Patients are randomized to 1 of 4 groups.

GROUP I: Patients watch an educational video about Mohs surgery before their surgery, a video about wound care after the surgery and receive text messages about wound care on days 1-5 after the surgery. Patients also receive instructions to reduce movement and use a Fitbit activity tracker. Beginning 48 hours after surgery, patients are instructed to apply petroleum jelly twice daily (BID) to the wound area.

GROUP II: Patients watch an educational video about Mohs surgery before their surgery, an educational video about wound care after the surgery and receive instructions to reduce movement and use a Fitbit activity tracker. Beginning 48 hours after surgery, patients apply petroleum jelly BID to the wound area.

GROUP III: Patients receive text messages about wound care on days 1-5 after the surgery and receive instructions to reduce movement and use a Fitbit activity tracker. Beginning 48 hours after surgery, patients are also instructed to apply petroleum jelly BID to the wound are.

GROUP IV: Patients receive no video or text messages. Patients receive instructions to reduce movement and use a Fitbit activity tracker. Beginning 48 hours after surgery, patients are also instructed to apply petroleum jelly BID to the wound area.

After completion of study, patients are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* The patient is undergoing Mohs surgery
* Subject is capable of understanding and willing to provide a signed and dated written voluntary informed consent before any protocol specific procedures are performed
* The subject is able to complete the study and comply with study instructions, including attending all study visits
* The patient has a cell phone capable of receiving text messages

Exclusion Criteria:

* The patient is not indicated for Mohs surgery
* Inability to complete all study-related visits
* Non-English speaking patients
* The patient cannot receive text messages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety score | Before surgery
  The preoperative anxiety scores of patients randomized to receive or not receive the educational video will be compared using a t-test or appropriate non-parametric test (Wilcoxon Rank Sum or Sign test) based on the distribution of the scores.
Patient knowledge score | Up to 1 week after completion of study
  Patient knowledge scores of patients randomized to receive or not receive the educational video will be compared using a t-test or appropriate non-parametric test (Wilcoxon Rank Sum or Sign test) based on the distribution of the scores.
Medication adherence | Up to 1 week after completion of study
  The mean number of times the medication was applied will be compared for the three intervention groups versus the control group.

SECONDARY OUTCOMES:
Patient satisfaction score | Up to 1 week after completion of study
  Patient satisfaction scores across the four randomization groups will be compared using analysis of variance (ANOVA) methods.
Mobility adherence as measured by Fitbit monitor | Up to 1 week after completion of study
  Compare the average number of steps taken each day between groups and the cumulative number of steps taken over the whole week using ANOVA methods. Percentage of patients with average daily activity below 2500 steps will be compared using the Chi-Squared or Fisher's Exact test. All three intervention groups will be compared to the control group.
Incidence of adverse events | Up to 1 week after completion of study
  The proportion of patients reporting adverse events will be compared using chi-squared tests or Fisher's exact tests, depending on the expected frequency of events. Comparisons will be made for those given versus not given the surgery education mobile app and then for those given versus not given text messages. To look at all four groups independently, a global statistic will be initially calculated. If significant, comparisons between the four groups will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pearce, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States